CLINICAL TRIAL: NCT04482205
Title: Covid -19 Pandemic: Economic Burden on Patients Operated for Traumatic Close Fractures in Musculoskeletal Service Line of a Tertiary Care Hospital
Brief Title: Covid -19 Pandemic: Economic Burden on Patients Operated for Traumatic Close Fractures
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, shah fahad, Resident, Aga Khan University
Other Study IDs: akupde
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Economic Burden
Keywords: economic burden, covid-19 pandemic
MeSH Terms: conditions — Financial Stress; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- precovid group: those who were operated from fJanuary first to March 15
- covid: those operated from March 16, to May 31, 2020

SUMMARY:
Covid-19 has adversely impacted the health care organizations by over burdening with Covid patients and suspending the elective surgeries and clinics A single center retrospective study was conducted to quantify losses due to postponement of elective surgeries and extra cost for procurement of PPEs. The secondary objective was to see the effect of Covid -19 on the total costs of inpatient care during Covid era.

DETAILED DESCRIPTION:
Covid-19 has impacted adversely the economy of Pakistan that has already poor and challenged socioeconomic conditions This is a single hospital retrospective cross sectional study conducted to quantify losses due postponement of elective surgeries and procurement of PPEs and see the effect of Covid -19 on the total costs of inpatient care during Covid era.

We included all the patients admitted in orthopedic section for operative intervention of fractures and elective procedures from January 1, 2020 to May 31, 2020. We divided this period into two halves; the first half was from January first to March 15 named as PreCovid Era and second half was from March 16, to May 31, 2020, termed as Covid Era. The total number of trauma procedures and elective procedures were compared in both eras. We compared six procedures each from upper and lower limit for cost analysis and length of stay. We also analyzed the extra cost for procurement of PPEs.

ELIGIBILITY:
Inclusion Criteria:

* All the patients admitted in orthopedic section for operative intervention of fractures and elective procedures from January 1, 2020 to May 31, 2020.

Exclusion Criteria:

* Patients presenting with other bone morbidities that did not require surgical interventions including rickets, osteomalacia, osteogenesis imperfecta, marble bone disease (osteopetrosis), Paget disease of bone, and fibrous dysplasia, patients with incomplete medical records were excluded from the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted for operative intervention of fractures management and elective procedures for tumour, degenerative disease, sport related injuries
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
the effect of Covid -19 on the total costs of inpatient care | 5 months
  the effect of Covid -19 on the total costs of inpatient care during Covid era

SECONDARY OUTCOMES:
drop in the collective revenue generated in covid era | 5 months
  to quantify drop in the collective revenue generated in covid era

CONTACTS AND LOCATIONS:
Overall Officials: Pervaiz Hashmi, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan